CLINICAL TRIAL: NCT03860038
Title: A Phase 2, Multi-center, Single-arm Study of TJ202 Combined With Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma Who Received at Least 2 Prior Lines of Treatment
Brief Title: TJ202 Combined With Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ202001MMY201
Record Dates: First submitted 2019-01-15; First posted 2019-03-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma in Relapse; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJ202 (Experimental)
  Interventions: Drug: TJ202 and Dexamethasone

INTERVENTIONS:
Drug: TJ202 and Dexamethasone — one dose of TJ202 16 mg/kg or an adjusted dose will be administered on Day 1 and Day 4 of Week 1, then every week from Week 2 to Week 12, then every 2 weeks from Week 13 to Week 24 and then every 4 weeks thereafter, until the subjects experience an onset of endpoint events like intolerance or PD. DEX 40 mg will be administered on Day 1 and Day 4 of Week 1, respectively and then 40mg weekly thereafter.

SUMMARY:
This trial is a multi-center, single-arm phase 2 study to evaluate the efficacy and safety of TJ202 combined with dexamethasone in subjects with relapsed or refractory multiple myeloma (RRMM) who received at least 2 prior lines of treatment.

DETAILED DESCRIPTION:
A total of 82 subjects with relapsed or refractory multiple myeloma (RRMM) who have received at least 2 prior lines of treatment will be enrolled in this study. Prior lines of treatment must include a proteasome inhibitor (PI) and an immunomodulator (IMiD). All subjects will receive TJ202 and dexamethasone (DEX) in the study. The treatment will continue until endpoint events such as intolerance or progressive disease (PD).

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18, male or female;
2. Subject must have had documented MM;
3. At screening phase, subject must have measurable disease;
4. Subject is in a state of progressive disease (PD);
5. Subject must have life expectancy of no less than 6 months;
6. Subject must have an ECOG (Eastern Cooperative Oncology Group) performance status score of 0~2;

Exclusion criteria:

1. Subject has received anti-CD38 monoclonal antibody treatment previously;
2. Subject has received CAR-T cell therapy previously;
3. Subject has previously received allogenic stem cell transplant, or subject has received autologous stem cell transplant within 3 months before administration of the study agent;
4. Primary refractory multiple myeloma (subject failed to generate any minimal response or any degree of response to any therapy);
5. Subject has received anti-myeloma treatment (radiotherapy is excluded) within 4 weeks or 5 PK half-lives of the treatment, whichever longer, before the first study agent administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | end of study [ Time Frame: Approximately up to 2 years ]
  defined as the proportion of subjects achieving stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and partial response (PR)

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | end of study [ Time Frame: Approximately up to 2 years ]
Duration of response (DOR) | end of study [ Time Frame: Approximately up to 2 years ]
Time to progression (TTP) | end of study [ Time Frame: Approximately up to 2 years ]
Time to response (TTR) | end of study [ Time Frame: Approximately up to 2 years ]
Progression-free survival (PFS) | end of study [ Time Frame: Approximately up to 2 years ]
Overall survival (OS) | end of study [ Time Frame: Approximately up to 2 years ]

OTHER OUTCOMES:
minimal residual disease (MRD) assessment | end of study [ Time Frame: Approximately up to 2 years ]
  For subjects reaching CR and above, their bone marrow samples will be collected for exploratory minimal residual disease (MRD) assessment at the central laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Doctor, Principal Investigator — Institute of Hematology & Hospital of Blood Diseases CAMS&PUMC
Locations (18):
- China (17):
  - Beijing Chao-Yang Hospital,Capital medical university, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Nanfang Hospital of SMU, Guangzhou, Guandong
  - The second people's Hospital of Shenzhen, Shenzhen, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangzhou
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The first Bethune hospital of Jilin University, Changchun, Jilin
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - National Taiwan University Hospital, Taiwan, Taiwan
  - Tri-Service General Hospital, Taiwan, Taiwan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital，affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, College of Medicine,Zhejiang University, Hangzhou, Zhejiang
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No